CLINICAL TRIAL: NCT06873646
Title: Wound Dressing Patch with Kelulut Honey-Infused Alginate (Tri-Gnate Alginate) for Effective Wound Care Management
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mohd Khairul Zul Hasymi Firdaus (Other)
Collaborators: Ministry of Higher Education, Malaysia (Other)
Responsible Party: Sponsor-Investigator, Mohd Khairul Zul Hasymi Firdaus, Principal Investigator, Prince of Songkla University
Organization: Prince of Songkla University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tri-Gnate Study
Record Dates: First submitted 2025-03-03; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — dermacyn

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tri-Gnate Alginate Dressing (Experimental)
  Interventions: Combination Product: Tri-Gnate Alginate Dressing
- Dressing product from Manuka honey (Active Comparator)
  Interventions: Combination Product: Dressing product from Manuka honey
- Bactigras + Dermcyn (Placebo Comparator)
  Interventions: Combination Product: Bactigras + Dermacyn

INTERVENTIONS:
Combination Product: Tri-Gnate Alginate Dressing — Patient will receive dressing product (Tri-Gnate Alginate) for the management of wound. The product will be put on every alternate day. Wound condition will be monitored from T0 - T6.
  Arms: Tri-Gnate Alginate Dressing
Combination Product: Dressing product from Manuka honey — Patient will receive other type of dressing product (Manuka honey product) for the management of wound. The product will be put on every alternate day. Wound condition will be monitored from T0 - T6.
  Arms: Dressing product from Manuka honey
Combination Product: Bactigras + Dermacyn — Patient will receive standard dressing product (bactigras + dermacyn) for the management of wound. The product will be changed everyday. Wound condition will be monitored from T0 - T6 on alternate day basis.
  Arms: Bactigras + Dermcyn

SUMMARY:
The main aim of this study to effectiveness of dressing patch with Kelulut honey (Tri-Gnate Alginate) in promoting wound healing compared to conventional treatments (standard wound dressing + bactigras) and other types of medicinal honey based product (Manuka honey product). Tri-Gnate alginate is a product produced by researcher team which upgraded from raw honey into a dressing patch. 110 patients with diabetic foot ulcers is expected to enrol in this program. The patients will be assigned randomly into 3 groups namely as Group 1 - patient that will receive Tri-Gnate alginate product in their dressing, Group 2 - patient will receive Manuka honey patch product and group 3 - the patient will receive standard care (bactigras dressing + dermacyn). Prior to the applying of these dressing treatment, all the patient will receive Maggot Debridement Therapy (MDT) to ensure the wound is clean. Patient's wound condition will be monitored 7 times (T0 - T6) on alternate day basis for healing improvement.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above.
2. present with sloughly diabetes-based foot ulcer
3. Has diabetic foot ulcers more than 2 weeks, less than 1 year.
4. HbA1c reading than 9.0
5. Ankle-brachial index pressure (ABPI) should > 0.8
6. No more than 1 diabetic foot ulcer per foot.
7. no known allergy to honey of bee products
8. keen on both honey and maggot debridement therapy (MDT)
9. DFU classification: Wagner Grade 2, 3
10. Amputation possibly deferred

Exclusion Criteria:

1. patient in critical state.
2. patient in confuse state.
3. patient do not understand Malay or English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Wound Size Reduction | Day1 - Day 14
  Wound size reduction will be measured and jot down into data collection document. The wound condition will be measured 7 times at T0 (baseline) until T6. The wound assessment camera software will be used to measure the size of the wound (in cm2). The measurement will be carried out every alternate day. The mean score reduction of wound size (in cm2) will be used to monitor the wound condition.
Time to healing | Day1 - Day 14
  Time to healing will be measured based on the progress of the wound healing according to the mean of days taken. The healing progress will be monitored T0 as baseline until T6 at Day 14.
Patient reported pain | Day1 - Day 14
  The patient reported pain will be measured by using numerical scale from 0 (no pain) to 10 (severe pain). The pain will be assessed before the changes of new dressing done. The pain will be monitored from baseline (T0) until Day 14 (T6). Mean score of pain will be used to describe the pain present.

SECONDARY OUTCOMES:
Fasting blood sugar (FBS) | Day1 - Day 14
  A 2-3 ml of blood will be extracted from the patient. The blood will be sent to laboratory for FBS testing. The FBS value should be within 4.4 to 7.0 mmol/L. The mean value of FBS will used to monitored the blood sugar control within the patient. Higher value of FBS showed that patient has no control of the sugar. FBS will be measured on the similar day of the changing of the dressing (T0 - T6).
Complete blood counts (CBC) | Day1 - Day 14
  A 2-3 ml of blood will be extracted from the patient. The blood will be sent to laboratory for CBC testing. In the CBC testing there are few components that really important and relevant to this study which are WBC, Neutrophil, lymphocyte, monocyte, eosinophil and basophil. The CBC value should be as follow: White blood cell (WBC), normal range (x10^9/L) is 2.79 - 8.09, Neutrophil (x10^9/L) is 0.91-4.61, lymphocyte (x10^9/L) is 1.12 - 3.15, monocytes (x10^9/L) is 0.23 - 0.72, eosinophil (x10^9/L) is 0.03 - 0.37 and basophil (x10^9/L) is 0.002 - 0.058. Higher counts of the stated components than normal range showed that the patient is possibly having infection. CBC will be measured on the similar day of the changing of the dressing (T0 - T6).

CONTACTS AND LOCATIONS:
Locations (1):
- IIUM Medical Centre, Kuantan, Pahang, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
IPD might not be shared since we are required to not disclose any patient's data by our ethical committee clearance.